CLINICAL TRIAL: NCT00520780
Title: A Randomised Double-blind Controlled Phase III Study to Compare the Efficacy and Safety of Intravenous Iron Carboxymaltose (Ferinject®) With Placebo in Patients With Chronic Heart Failure and Iron Deficiency
Brief Title: Ferinject® Assessment in Patients With Iron Deficiency and Chronic Heart Failure (FAIR-HF)
Acronym: FAIR-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Collaborators: Syneos Health (Other); ClinStar, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FER-CARS-02
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2010-03

CONDITIONS: Chronic Heart Failure; Iron Deficiency; Iron Deficiency Anemia; Anaemia
Keywords: Chronic Heart Failure; Iron deficiency; Iron deficiency anaemia; Anaemia; Heart disease
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency; Anemia; Heart Diseases | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Ferinject ® (Ferric carboxymaltose)
- 2 (Placebo Comparator)
  Interventions: Drug: Normal saline (0.9%)

INTERVENTIONS:
Drug: Ferinject ® (Ferric carboxymaltose) — Ferinject® will be administered in doses of 200 mg (4 mL) weekly up to iron repletion (correction phase of variable duration depending on individual iron deficit). The calculated dose will be rounded to the next 100 mg iron, i.e. the final dose may be 100 mg iron depending on the individual iron deficit.
  After the correction phase, Ferinject® will be given monthly in doses of 200 mg until the 24th week (maintenance phase).
  Arms: 1
Drug: Normal saline (0.9%) — During the correction phase, patients will receive the number of normal saline injections (4 mL weekly) corresponding to the calculated total iron dose needed according to the individual iron deficit. During the maintenance phase, placebo patients will receive 4 mL normal saline monthly.
  Arms: 2

SUMMARY:
This study is designed to evaluate the efficacy of Ferinject® in improving symptoms of CHF in patients with iron deficiency. Analyses will focus both on subjective and objective measures. Furthermore, the tolerability and safety of Ferinject® treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* In New York Heart Association (NYHA) II-III functional class due to stable symptomatic chronic heart failure (CHF)
* Left ventricular ejection fraction (LVEF) 40% or lower for patients in NYHA II and 45% or lower in NYHA III
* Screening haemoglobin (Hb) at least 9.5 g/dL but below or equal to 13.5 g/dL (average of 2 haemoglobin concentrations)
* Screening ferritin below 100 µg/L, or below 300 µg/L when transferrin saturation (TSAT) is below 20%

Exclusion Criteria:

* History of acquired iron overload.
* Known active infection, clinically significant bleeding, active malignancy.
* Chronic liver disease and/or screening alanine transaminase (ALT) or aspartate transaminase (AST)
* Anaemia due to reasons other than iron deficiency
* Immunosuppressive therapy or renal dialysis (current or planned within the next 6 months).
* History of erythropoietin, i.v. or oral iron therapy, and blood transfusion in previous 12 weeks and/or such therapy planned within the next 6 months.
* Unstable angina pectoris as judged by the investigator, clinically significant uncorrected valvular disease or left ventricular outflow obstruction, obstructive cardiomyopathy, poorly controlled fast atrial fibrillation or flutter, poorly controlled symptomatic brady- or tachyarrhythmias.
* Acute myocardial infarction or acute coronary syndrome, transient ischaemic attack or stroke within the last 3 months.
* Coronary-artery bypass graft, percutaneous intervention (e.g. cardiac, cerebrovascular, aortic; diagnostic catheters are allowed) or major surgery, including thoracic and cardiac surgery, within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2007-04; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Self-reported patient global assessment (PGA) and NYHA functional status 24 weeks after initiation of therapy | 24 weeks

SECONDARY OUTCOMES:
Key secondary objectives (efficacy): Exercise tolerance (6-minute walk test distance). Further secondary objectives(efficacy): Health related quality of life, resource use and costs associated with the treatment, safety and tolerability | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Poole-Wilson, MD FRCP, Principal Investigator — National Heart and Lung Institute. Faculty of Medicine. Imperial College London. Dovehouse Street, London SW3 6LY, UK
Locations (48):
- Research Sites, Buenos Aires, Argentina
- Germany (9):
  - Research Site, Bad Nauheim
  - Research Site, Berlin
  - Research Site, Göttingen
  - Research Site, Hanover
  - Research Sites, Heidelberg
  - Research Site, Herford
  - Research Site, Herne
  - Research Site, Kiel
  - Research Site, München
- Greece (2):
  - Research Site, Athens
  - Research Site, Heraklion
- Italy (4):
  - Research Site, Ascoli Piceno
  - Research Site, Pavia
  - Research Site, Rome
  - Research Site, Vicenza
- Research Site, Stavanger, Norway
- Poland (11):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Opole
  - Research Site, Piotrkow Trybunalski
  - Research Site, Siedlce
  - Research Site, Torun
  - Research Sites, Warsaw
  - Research Site, Wałbrzych
  - Research Site, Wroclaw
  - Research Site, Włocławek
  - Research Site, Zabrze
- Romania (4):
  - Research Site, Brasov
  - Research Sites, Bucharest
  - Reserach Site, Craiova
  - Research Sites, Târgu Mureş
- Russia (3):
  - Reserach Sites, Moscow
  - Resarch Sites, Saint Petersburg
  - Research Sites, Veliky Novgorod
- Spain (5):
  - Research Site, Alicante
  - Research Sites, Barcelona
  - Research Site, Bilbao
  - Research Site, Madrid
  - Research Site, Valencia
- Ukraine (8):
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Sites, Kiev
  - Research Site, Lviv
  - Research Site, Mykolayiv
  - Research Site, Odesa
  - Research Site, Zaporizhzhya

REFERENCES:
- [Derived] Anker SD, Comin Colet J, Filippatos G, Willenheimer R, Dickstein K, Drexler H, Luscher TF, Bart B, Banasiak W, Niegowska J, Kirwan BA, Mori C, von Eisenhart Rothe B, Pocock SJ, Poole-Wilson PA, Ponikowski P; FAIR-HF Trial Investigators. Ferric carboxymaltose in patients with heart failure and iron deficiency. N Engl J Med. 2009 Dec 17;361(25):2436-48. doi: 10.1056/NEJMoa0908355. Epub 2009 Nov 17. PMID 19920054
- [Derived] Anker SD, Colet JC, Filippatos G, Willenheimer R, Dickstein K, Drexler H, Luscher TF, Mori C, von Eisenhart Rothe B, Pocock S, Poole-Wilson PA, Ponikowski P; FAIR-HF committees and investigators. Rationale and design of Ferinject assessment in patients with IRon deficiency and chronic Heart Failure (FAIR-HF) study: a randomized, placebo-controlled study of intravenous iron supplementation in patients with and without anaemia. Eur J Heart Fail. 2009 Nov;11(11):1084-91. doi: 10.1093/eurjhf/hfp140. PMID 19875408